CLINICAL TRIAL: NCT07057622
Title: Compare the Safety and Efficacy of 177Lu-DOTATATE and Octreotide LAR in Unresectable or Metastatic, Progressive, Well-differentiated(G1 and G2) and SSTR-positive Adult GEP-NEN
Brief Title: A Phase III Clinical Study to Compare the Safety and Efficacy of 177Lu-DOTATATE Injection and Long-acting Oxytrexine in Adult Patients With NETs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HTA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YZGK-ZLYT-2023-Ⅲ-Lu
Record Dates: First submitted 2024-09-13; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: NETS Ga68 Lu177
MeSH Terms: interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 177Lu-DOTATATE Injection (Experimental): Subjects in the test group are treated with 177Lu-DOTATATE injection, 7.4GBq±0.74GBq (200mCi±20mCi)/cycle, once every 8 to 12 weeks, 4 times in total.
  Interventions: Drug: 177Lu-DOTATATE injection
- Octreotide LAR (Active Comparator): Subjects in the treatment group are treated with 60mg of long-acting octreotide once every 4 weeks±3 days.
  Interventions: Drug: Octreotide LAR (Long-acting release)

INTERVENTIONS:
Drug: 177Lu-DOTATATE injection — The eligible subjects who participate in 177Lu study are randomly assigned 1:1 to either the test group or the control group to receive treatment. Subjects in the test group are treated with 177Lu-DOTATATE injection, 7.4GBq±0.74GBq (200mCi±20mCi)/cycle, once every 8 to 12 weeks, 4 times in total.
  Arms: 177Lu-DOTATATE Injection
Drug: Octreotide LAR (Long-acting release) — The eligible subjects who participate in 177Lu study are randomly assigned 1:1 to either the test group or the control group to receive treatment. Subjects in the treatment group are treated with 60mg of long-acting octreotide once every 4 weeks±3 days.
  Arms: Octreotide LAR

SUMMARY:
The study is to evaluate the sstr antagonists, 68Ga-DOTATATE and 177Lu-DOTATATE,as a pair of diagnostic/therapeuticradiopharmaceuticals(theranostics)in patients with NETS

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document;
2. Age ≥18 years ;
3. Low-and medium-grade ( G1 or G2) unresectable locally advanced or metastaticgastrointestinalneuroendocrine tumors(GEP-NETs)confirmed by histopatholog in the central laboratory,and those who had previously progressed after standard-dose somatostatin analogue(SSA)treatment;
4. Somatostatin receptor positive patients must be defined as all target lesions at baseline confirmed by PET/ CT examination of gallium [68Ga] dobutamine injection as somatostatin receptor positive(IRC confirmed);
5. There is at least one measurable lesion at baseline;
6. BaselineECOG score 0 or 1;
7. Adeguate organ and bone marrow function as defined below:

   a) bone marrow:Neutrophil count (ANC)≥1.5×109/L, platelet count ≥75×109/L,hemoglobin ≥80g/L,no blood transfusion or growth factor treatment within 14 days before randomization.(colony stimulating factor (CSF), colony stimulating factor (CSF),Erythropoietin(EPO),etc.); b) Liver function:aspartate aminotransferase(AST)and alanine aminotransferase(ALT)≤2.5 ULN; total bilirubin( TBIL ) ≤1.5 × ULN; c ) Renal function : serum creatinine ≤150μmol/ L or 1.7mg / dL, or creatinine clearance rate (CLcr)≥50mL/min calculated by Cockroft Gault method; d) Baseline left ventricular ejection fraction (LVEF)≥50 % measured by multi-gate circuit controlled acquisition(MUGA) or echocardiography(ECHO); e ) Coagulation function: international normalized ratio(INR)≤1.5 ×ULN,activated partial thromboplastin time(APTT ) ≤1.5 × ULN ; f) Serum albumin > 3.0g/ dL.
8. Subjects with childbearing potential voluntarily use effective contraceptive methods,such as condoms, oral or injectable contraceptives, intrauterine devices, etc, during treatment and within 4 months (men) or 7months(women)after the last use of the investigational drug.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) antibody positive;
2. Hepatitis B virus (HBV) surface antigen (HBsAg) is positive and HBV-DNA is positive (≥the upper limit of detection), or hepatitis C virus (HCV) antibody (HCV-Ab) is positive and HCV-RNA is positive (≥the upper limit of detection));
3. Pregnant or lactating women;
4. Received peptide receptor radionuclide therapy (PRRT) before randomization;
5. Received Octreotide LAR treatment with a dose intensity >30 mg/3-4 weeks (increased dose or frequency) within 12 weeks before randomization;
6. Subjects who are receiving short-acting octreotide treatment cannot stop short-acting octreotide within 24 hours before and 24 hours after administration of 177Lu-DOTATATE or subjects who are receiving Octreotide LAR treatment cannot stop Octreotide LAR within 4 weeks before administration of 177Lu-DOTATATE;
7. Have received systemic anti-tumor treatments such as targeted therapy, immunotherapy,anti-tumor Chinese medicine treatment, chemotherapy,etc.within 4 weeks before randomization;
8. Participated in other drug clinical trials and received corresponding experimental drugs within 4 weeks before randomization, except for the PET/CT study of the diagnostic drug68Ga-DOTATATE injection initiated by the sponsor of this trial;
9. Received the following treatments within 12 weeks before randomization,including but not limited to surgery (except biopsy),radical radiotherapy,hepatic artery interventional embolization,cryoablation or radiofrequency ablation of liver metastases;
10. Received palliative radiotherapy for bone metastases within 2 weeks before randomization;
11. The toxicity of previous anti-tumor treatment has not recovered to s grade 1 level (except for hair loss and neurotoxicity);
12. Known brain metastasis (except those who have received treatment and been stable for at least 24 weeks before randomization);
13. Severe cardiac insufficiency,including congestive heart failure 2 grade 2 (New York Heart Association classification), myocardial infarction, stroke or transient ischemic attack (TIA) history within 6 months before enrollment; 14.History of ventricular tachycardia or torsade de pointes.Any clinically important abnormality in resting ECG rhythm, conduction,or morphology, such as QTcF >450 msec in men or QTcF>470 msec in women, the presence of complete left bundle branch block or third-degree atrioventricular block;

15. Pulmonary embolism or deep vein thrombosis occurred within 3months before randomization; 16.Uncontrolled hypertension(e.g.systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)and uncontrolled diabetes ( baseline fasting blood glucose >8.9 mmol/ L or glycosylated hemoglobin(HbA1C)>6.5%); 17.There were uncontrolled active bacterial, viral,fungal,rickettsial or parasitic infections requiring intravenous anti-infective therapy within the first 2 weeks of randomization; 18.There were concurrent malignant tumors within the first 5 years of enrollment (except for fully treated cervical carcinoma in situ,localized skin squamous cell carcinoma,basal cell carcinoma, prostate cancer without anti-tumor treatment,thyroid cancer,breast ductal carcinoma in situ, and urothelial carcinoma below T1); 19. Known allergies to 68Ga-DOTATATE injection or 177Lu-DOTATATE injection or Octreotide LAR components and theirexcipients; 20. Any other disease or mental state that is not under control and may affect the completion of the study (including poor compliance) or is not suitable for the use of experimental drugs; 21.According to the patient 's disease characteristics,the researchers believe that other treatment options (such as chemotherapy,targeted therapy) are more suitable for patients than the treatment provided in the study,that is,the experimental drugs are not the best therapeutic drugs in clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2027-02-24 (Estimated)

PRIMARY OUTCOMES:
Compare the 18-month PFS rate of NET patients between 177Lu-DOTATATE Injection and long-acting octreotide | 18 months from enrollment to PFS
  Compare the 18-month PFS rate of NET patients between 177Lu-DOTATATE Injection and long-acting octreotide

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided